CLINICAL TRIAL: NCT03992248
Title: Effect of Time Restricted Feeding on Hepatic Glycogen Depletion and Insulin Sensitivity in Adults With Type 2 Diabetes
Brief Title: Effect of Eating Within a Limited Time on Sugar Sensitivity and Liver Sugar Stores of People With Type 2 Diabetes.
Acronym: TRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NL67610068
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: TRF; Hepatic glycogen; Type 2 diabetes; Insulin sensitivity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Randomised controlled cross-over design with two 3-week arms and a 4-week wash-out period.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of this study, it is not possible to mask the intervention effect for the investigator or the participant. During randomisation, the intervention arms will be coded with 1 and 2 and the independent researcher will be unaware which intervention is assigned to which letter. With this approach, concealed allocation will be guaranteed. Additionally, the person in charge with the data quality check and the data analyses will be blinded for the interventions using this same randomisation codes to generate unbiased results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time Restricted Feeding (Experimental): Participants are instructed to eat within a limited time frame during the day. They are also instructed to keep record of their eating and sleeping record with eat- and sleep diaries.
  Interventions: Behavioral: Time restricted feeding
- Control (Other): Participants are instructed to spread their habitual food intake over at least 14hrs per day. They are also instructed to keep record of their eating and sleeping record with eat- and sleep diaries.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Time restricted feeding — Eating within a time frame of 10hrs during the day. Outside of this time frame, participants need to refrain from food and energy containing drinks.
  Arms: Time Restricted Feeding
Behavioral: Control — Eating for at least 14hrs per day.
  Arms: Control

SUMMARY:
Modern life is characterized by a 24-hour lifestyle in which food intake is no longer restricted to daytime. As a result, people nowadays tend to eat throughout the day. When food is being consumed the energy is both used and stored for later use. Eating for a prolonged period of time makes it unnecessary for the body to use its energy storage. It is hypothesized that the decreased use of energy stores has detrimental effects on our sugar balance, mainly on insulin sensitivity. Conversely, eating within a limited period during the day could improve insulin sensitivity in people with type 2 diabetes by an increased use of energy reserves, specifically liver sugar stores. Therefore, this study examines the effect of eating within a limited time frame during the day on insulin sensitivity and liver sugar stores of people with type 2 diabetes.

DETAILED DESCRIPTION:
Modern life is characterized by a 24-hour lifestyle in which food intake is no longer restricted to daytime. Interestingly, the majority of people spread their food intake over ~15 hours per day. This implies that most people experience a relatively short post-absorptive (fasting) state during night time. Normally, the body relies heavily on hepatic glycogen content to provide glucose and energy during the night, and glycogen stores will therefore decrease over night. In the morning, ingested carbohydrates will be taken up rapidly to replenish glycogen stores. It is hypothesized that in people with type 2 diabetes mellitus (T2DM) hepatic glycogen stores may not fully deplete overnight and that restricting food to a shorter period of time during the day will lead to a reduction of hepatic glycogen stores, and thereby improve whole-body insulin sensitivity at the beginning of the day. Therefore, the aim of this study is to investigate if time restricted feeding (TRF) leads to a reduction in overnight-fasted hepatic glycogen stores and improvement in insulin sensitivity in adults with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Caucasian
* Non-insulin treated type 2 diabetes,
* BMI: >25 kg/m2
* Regular sleeping time (normally 7 - 9 hrs daily)
* Habitual bedtime at 11 PM plus/minus 2 hours

Exclusion Criteria:

* Not being able to adhere to a restricted feeding schedule
* Uncontrolled hypertension
* Active cardiovascular disease
* Insulin therapy
* Use of SGLT2 inhibitors
* BMI>38 kg/m2
* Engaged in programmed exercise for >3hrs per week
* Extreme early bird or extreme night person
* Heavily varying sleep-wake rhythm
* Shiftwork during last 3 months
* Smoking
* Contra-indication to MRI scanning
* Subjects who intend to donate blood during the intervention or subjects who have donated blood less than three months before the start of the intervention
* Subjects who do not want to be informed about unexpected medical findings during the screening/study, or do not wish that their physician is informed
* Unstable body weight (weight gain or loss >3kg in the last 3 months)
* Significant food allergies/intolerance (seriously hampering study meals)
* Participation in another biomedical study within 1 month before the first study visit, which would possibly hamper our study results
* Any other medical condition that will preclude the safe performance of the measurements

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2021-02-03 (Actual)

PRIMARY OUTCOMES:
Hepatic glycogen | Measurement performed after 3 weeks of intervention/control
  13C-Magnetic Resonance Spectrometry

SECONDARY OUTCOMES:
Insulin sensitivity | Measurement performed after 3 weeks of intervention/control
  Two-steps hyperinsulinaemic clamp

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schrauwen, Prof. Dr., Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Andriessen C, Fealy CE, Veelen A, van Beek SMM, Roumans KHM, Connell NJ, Mevenkamp J, Moonen-Kornips E, Havekes B, Schrauwen-Hinderling VB, Hoeks J, Schrauwen P. Three weeks of time-restricted eating improves glucose homeostasis in adults with type 2 diabetes but does not improve insulin sensitivity: a randomised crossover trial. Diabetologia. 2022 Oct;65(10):1710-1720. doi: 10.1007/s00125-022-05752-z. Epub 2022 Jul 25. PMID 35871650